CLINICAL TRIAL: NCT03850938
Title: Comparison of Kyphoplasty With and Without Rotary Cutter Subacute Osteoporotic Vertebral Fractures
Brief Title: Percutaneous Kyphoplasty Using Rotary Cutter in Osteoporotic Vertebral Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Li Min (Other)
Responsible Party: Sponsor-Investigator, Li Min, Vice Director, Jinan Military General Hospital
Organization: Jinan Military General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 960HP20190012
Record Dates: First submitted 2019-02-20; First posted 2019-02-22 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Spine Fracture
Keywords: fractures, compression; back pain; bone cements; kyphoplasty
MeSH Terms: conditions — Spinal Fractures; Fractures, Compression; Back Pain | interventions — Kyphoplasty

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Kyphoplasty (Experimental): The balloon is first placed into the fractured vertebra and inflated with contrast agent for height restoration. Then, the cement is injected into the cavity created by the balloon.
  Interventions: Device: Conventional Kyphoplasty
- Kyphoplasty with Rotary Cutter (Active Comparator): The balloon is first placed into the fractured vertebra and inflated with contrast agent for height restoration, which may induce a cavity with barriers pushed by balloon dilatation. Then, the structure of the cavity is destroyed by a rotary cutter. Finally, the cement is injected, which may effectively interdigitates with the healthy cancellous bone.
  Interventions: Device: Kyphoplasty with Rotary Cutter

INTERVENTIONS:
Device: Conventional Kyphoplasty — The cement is injected into the cavity created by PKP. The diffusion of cement can be interfered by closely barriers formed by surrounding cancellous bones.
  Other Names: Conventional PKP
  Arms: Conventional Kyphoplasty
Device: Kyphoplasty with Rotary Cutter — The rotary cutter is applied before cement injection to destroy the structure around the cavity created by inflated balloon. Then, the rotary cutter will make the bone cement to support a wider range and to blend with the surrounding cancellous bones more densely.
  Other Names: PKP with Rotary Cutter
  Arms: Kyphoplasty with Rotary Cutter

SUMMARY:
Kyphoplasty(PKP) is performed under general anaesthesia in patients with osteoporotic vertebral compression fracture. The balloon is first placed into the fractured vertebra and inflated with contrast agent for height restoration. Then, the cement is injected into the cavity created by the balloon. As the diffusion of cement can be interfered by closely barriers formed by surrounding cancellous bones, refractures are often found in patients with conventional PKP. Furthermore, the loss of restored height of surgical vertebrae due to refracture in PKP. The investigators will applied a rotary cutter to destroy the structure of the cavity created by the balloon. Finally, the cement is injected, which may effectively interdigitates with the surrounding cancellous bone.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is able to undergo the vertebroplasty or balloon kyphoplasty procedure
2. Patient has read and sign the informed consent
3. Male or female, 50 years or older
4. Compressive and burst vertebral body fractures without any neurological deficit.
5. Persistent pain despite medical treatment according to VAS ≥ 5 or a last resort to morphine treatment

Exclusion Criteria:

1. Neurological signs related to the vertebral fracture to treat
2. Unmanageable bleeding disorder
3. History of surgical or percutaneous spine treatment except simple discectomy at a single or multiple vertebral levels with no residual pain.
4. Known allergy to bone cement
5. Local or generalized infection
6. Improvement of the symptoms of the patient with conservative management

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Back pain: Visual analogue scales system | up to 2 years
  Measuring and comparing the post-operative back pain via Visual analogue scales system

SECONDARY OUTCOMES:
Refracture | up to 2 years
  Number of new vertebral fractures documented radiologically
Kyphotic angle and global thoracic and lumbar angulations | up to 2 years
The patterns of cement opacification | during the procedure of PKP
  The patterns of cement opacification were classified as solid patterns (cement forms a mass), trabecular patterns (cement spread along the fine bone trabeculae), and mixed patterns (cement forms a mass with spreading along the fine bone trabeculae)
Height of the treated vertebral body | Preoperative, up to 2 years
  Follow-up of anterior, median and posterior height of the treated vertebral body, obtained by making an average of all measurements
Medico-economic follow-up | up to 2 years
  Cost of intervention; Cost of prescribed medicines; Cost of follow-up visits; Cost of subsequent hospitalization; Cost of complications.

CONTACTS AND LOCATIONS:
Locations (1):
- Min Li, Jinan, Shandong, China